CLINICAL TRIAL: NCT01039272
Title: Epstein-Barr Detection in Squamous Cell Carcinoma and Healthy Oral Mucosa
Brief Title: Epstein-Barr Detection in Oral Cancer
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Sponsor
Other Study IDs: upeclin/FOA-Unesp-03
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Oral Cancer
Keywords: oral cancer; EBV; PCR
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — paraffin-embedded tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- oral cancer: patients with oral squamous cell carcinoma
- control group: healthy patients without any oral pathology

SUMMARY:
The aim of this study is to analyze oral squamous cell carcinoma and healthy oral mucosa for the possible presence of Epstein-Barr virus (EBV).

DETAILED DESCRIPTION:
Epstein-Barr virus has been implicated in a range of malignant neoplasms, including in some studies, in the aetiology of oral squamous cell carcinoma but the influence of EBV in oral cancer remains unclear. This study will examine the prevalence of EBV infection in oral cancer by means of nested polymerase chain reaction.

ELIGIBILITY:
Inclusion Criteria:

* patients of Oral Cancer Centre - UNESP/Araçatuba - SP
* with oral squamous cell carcinoma

Exclusion Criteria:

* without oral squamous cell carcinoma

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: oral care clinic, community sample
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
presence of EBV | 1 hour
  Epstein-Barr virus has been implicated in a range of malignant neoplasms, including in some studies, in the aetiology of oral squamous cell carcinoma but the influence of EBV in oral cancer remains unclear. This study will examine the prevalence of EBV infection in oral cancer by means of nested polymerase chain reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Glauco Issamu I Miyahara, Professor, Principal Investigator — Department of Pathology and Propaedeutics, Sao Paulo State University, Unesp, Araçatuba/SP; Lívia T Arêde, student, Study Chair — Department of Pathology and Propaedeutics, Sao Paulo State University, Unesp, Araçatuba/SP
Locations (1):
- Department of Pathology and Propaedeutics, Sao Paulo State University, Unesp, Araçatuba/SP, Araçatuba, São Paulo, Brazil

REFERENCES:
- See also: School of Dentistry, Sao Paulo State University, Unesp, Araçatuba/SP — http://www.foa.unesp.br